CLINICAL TRIAL: NCT05285813
Title: A Phase II Study of Vibecotamab (XmAb14045) for MRD- Positive AML and MDS After Hypomethylating Agent Failure
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1124; NCI-2022-02215 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-03-08; First posted 2022-03-18 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: AML; MDS
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; Acetaminophen; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AML MRD cohort only (Experimental): Each study cycle is 28 days. Vibecotamab by vein (IV) over about 2 hours On Days 1, 3, 5, 8, 15 and 22 of Cycle 1 and then on Days 1, 8, 15 and 22 of Cycles 2-4.
  Interventions: Drug: Vibecotamab; Drug: Dexamethasone; Drug: Acetaminophen; Drug: Diphenhydramine
- MDS post-HMA failure cohort only (Experimental): Each study cycle is 28 days. Vibecotamab by vein (IV) over about 2 hours On Days 1, 3, 5, 8, 15 and 22 of Cycle 1 and then on Days 1, 8, 15 and 22 of Cycles 2-4.
  Interventions: Drug: Vibecotamab; Drug: Dexamethasone; Drug: Acetaminophen; Drug: Diphenhydramine

INTERVENTIONS:
Drug: Vibecotamab — Given by vein (IV)
  Other Names: XmAb14045
Drug: Dexamethasone — Given by vein (IV) over about 60 minutes before the dose
  Other Names: Decadron
Drug: Acetaminophen — Given by mouth (PO) about 30-60 minutes before the dose
  Other Names: TylenolÂ®; DorcolÂ®; Feverallâ"¢; PanadolÂ®; APAP; N-Acetyl-P-Aminophenol; Paracetamol; Ofirmevâ"¢
Drug: Diphenhydramine — Given by mouth (PO) or Given by vein (IV) about 30-60 minutes before the dose
  Other Names: BenadrylÂ®

SUMMARY:
This is a phase II single-center study to evaluate the safety and effectiveness of vibecotamab, a CD3-CD123 bispecific antibody, in patients with acute myeloid leukemia with persistent or recurrent measurable residual disease and in patients with myelodysplastic syndrome that has not responded to or relapsed after conventional therapy

DETAILED DESCRIPTION:
Primary Objectives:

* AML MRD cohort: To determine the MRD negativity rate after 4 cycles of vibecotamab in patients with AML with MRD
* MDS post-HMA cohort: To determine the response rate (defined as CR + marrow CR [mCR] + partial remission [PR] + hematologic improvement [HI]) after 4 cycles of vibecotamab in patients with MDS after HMA failure

Secondary Objectives:

* To assess other efficacy endpoints, including remission duration, duration of MRD response (AML MRD arm only), CR rate (MDS arm only), relapse-free survival, overall survival
* To assess the safety of vibecotamab in patients with AML with MRD and in patients with MDS post-HMA failure

Exploratory Objectives:

* To correlate clinical outcomes with CD123 expression
* To determine the CD123 expression in patients who relapse after vibecotamab therapy

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age
2. AML MRD cohort only: AML in first or second morphologic remission (defined as complete remission [CR], complete remission with incomplete hematologic recovery [CRi], or morphologic leukemia-free state [MLFS]) who have received a minimum prior therapy with at least 1 course of intensive intermediate to high-cytarabine-based chemotherapy or at least 2 courses of lower-intensity therapy (e.g. hypomethylating agent or low-dose cytarabine-based)
3. AML MRD cohort only: Persistent or recurrent MRD positivity detected by MFC at a level of ≥0.1%.
4. AML MRD cohort only: For patients who are MRD positive by MFC, residual leukemia must be positive for CD123 expression at a level of at least 20% (as assessed by clinical pathologist)
5. MDS post-HMA failure cohort only: MDS that is intermediate, high risk or very high risk by the Revised International Prognostic Scoring System (IPSS) or CMML-1 or CMML-2 who have not responded after at least 4 cycles of azacitidine and/or decitabine or who progressed or relapsed after azacitidine and/or decitabine, regardless of the number of cycles received
6. MDS post-HMA failure cohort only: Aberrant blasts must be positive for CD123 expression by MFC at a level of at least 20% (as assessed by clinical pathologist)
7. Performance status 2 (ECOG Scale).
8. Female patients of childbearing potential must agree to use a highly effective method of birth control during and for 4 weeks after the last dose of vibecotamab and must also refrain from oocyte donation during this time period. Women are considered to be of childbearing potential unless it is documented that they are over the age of 60 OR postmenopausal by history with no menses for 1 year and confirmed by follicle-stimulating hormone (using local reference ranges) OR have a history of hysterectomy and/or bilateral oophorectomy OR have a history of bilateral tubal ligation. Highly effective methods of birth control include hormonal birth control (oral, intravaginal, transdermal, implantable, or intrauterine), intrauterine devices, vasectomized partner, or any double-barrier methods (combination of male condom and spermicide with either cap, diaphragm, or sponge).
9. Male patients and their female partner of childbearing potential must agree to use highly effective contraception, as above, and refrain from donating sperm during the treatment period and for at least 4 weeks after the last dose of vibecotamab.
10. Signed informed consent

Exclusion Criteria:

1. Prior treatment with vibecotamab or anti-CD123-directed therapy.
2. Clinically significant organ dysfunction, defined as:

   1. AST or ALT >3x the upper limit of normal (ULN)
   2. Total bilirubin >1.5x the ULN, unless due to ongoing hemolysis or Gilbert's syndrome
   3. Creatinine clearance <30 mL/min
   4. Active Grade III-V cardiac failure as defined by the New York Heart Association Criteria.
3. Active serious infection not controlled by oral or intravenous antibiotics (e.g. persistent fever or lack of clinical improvement despite antimicrobial treatment).
4. Patients who are expected to be able to proceed with stem cell transplantation within the next 30 days
5. Known human immunodeficiency virus (HIV) with detectable viral load.
6. Known hepatitis B surface antigen seropositive or known or suspected active hepatitis C infection Note: Patients who have isolated positive hepatitis B core antibody (ie, in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Patients who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load.
7. Patients with a prior or concurrent malignancy whose natural history or treatment is not anticipated to interfere with the safety or efficacy assessment of the investigational regimen may be included only after discussion with the PI
8. Treatment with any antileukemic agents or chemotherapy agents in the last 7 days or 5 half-lives (whichever is sooner) before study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the MRD negativity rate after 4 cycles of vibecotamab in patients with AML with MRD | through study completion, an average of 1 year
To determine the response rate (defined as CR + marrow CR [mCR] + partial remission [PR] + hematologic improvement [HI]) after 4 cycles of vibecotamab in patients with MDS after HMA failure | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Short, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org